CLINICAL TRIAL: NCT02384512
Title: Azilect® In Wearing-Off (AIWO) Non-interventional Study on Efficacy and Tolerability of Rasagiline (1mg/d) add-on in Ambulatory Parkinson's Disease Patients With Wearing-off Symptoms Diagnosed by Wearing-off Questionnaire (WOQ-32)
Brief Title: Azilect® In Wearing-Off (AIWO)
Acronym: AIWO
Status: Completed | Type: Observational
Sponsor: Teva Pharma GmbH (Industry)
Collaborators: Anfomed GmbH (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Other Study IDs: TVP1012-CNS-40090
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; akinesia; Azilect®; Rasagiline; Combination therapy with L-dopa; Wearing-off Questionnaire-32; Quality of life; Daily practice
MeSH Terms: conditions — Parkinson Disease | interventions — rasagiline

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Azilect® — AZILECT® 1mg Tablets
  Other Names: Rasagiline

SUMMARY:
End-of-dose fluctuations e. g. wearing-off are defined as a recurrence of motor and non-motor Parkinson's Disease (PD) symptoms that precedes a scheduled dose and improves with the next dose of anti-parkinsonian medication. Azilect® is approved and recommended for therapy of wearing-off-/End-of-dose fluctuations and improves motor fluctuations significantly in combination therapy with L-dopa and other parkinsonian medication.

DETAILED DESCRIPTION:
The aim of the non-interventional study is to document efficacy and tolerability of rasagiline as a combination therapy in patients with wearing-off-/End-of-dose fluctuations and the effect of rasagiline on individual wearing-off symptoms, recognized by wearing-off questionnaire 32 (WOQ-32).

ELIGIBILITY:
Inclusion:

* idiopathic Parkinson's disease based on the UK Brain Bank criteria,
* Wearing-off / end-of-dose akinesia
* at least 18 years old,
* written consent to participate in the study.

Exclusion:

* contraindications according to the SmPC of Azilect®,
* treatment with Azilect® in the past 3 months and / or
* suffering from a relevant cognitive impairment and therefore neither understand the patient information, nor can give their consent to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients with Parkinson's disease in Germany
Sampling Method: Probability Sample
Enrollment: 261 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Wearing-off Questionnaire-32 (WOQ-32) | 12 weeks
  Alterations of 32 different wearing-off symptoms (Patient questionnaire)

SECONDARY OUTCOMES:
WHO-5 | 12 weeks
  Alterations of patient's Quality of life (patient questionnaire)
GI-I | 12 weeks
  Self-Assessment of global improvement (patient questionnaire)
Columbia University Rating Scale (CURS) | 12 weeks
  Alteration of PD symptoms (physician rated questionnaires)
Clinical global impression improvement (CGI-I) | 12 weeks
  (physician rated questionnaires)
Percentage of participants with adverse events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Expert, MD, Study Director — Paracelsus Elena Klinik
Locations (140):
- Germany (140):
  - Teva Investigational Sites, Aalen
  - Teva Investigational Sites, Achim
  - Teva Investigational Sites, Altenburg
  - Teva Investigational Sites, Altenholz
  - Teva Investigational Sites, Alzenau in Unterfranken
  - Teva Investigational Sites, Apolda
  - Teva Investigational Sites, Aschaffenburg
  - Teva Investigational Sites, Bad Honnef
  - Teva Investigational Sites, Bad Kissingen
  - Teva Investigational Sites, Bad Mergentheim
  - Teva Investigational Sites, Bad Schwartau
  - Teva Investigational Sites, Bad Waldsee
  - Teva Investigational Sites, Bad Wörishofen
  - Teva Investigational Sites, Bensheim
  - Teva Investigational Sites, Bergisch Gladbach
  - Teva Investigational Sites, Berlin
  - Teva Investigational Sites, Bernburg
  - Teva Investigational Sites, Bielefeld
  - Teva Investigational Sites, Bochum
  - Teva Investigational Sites, Bockhorn
  - Teva Investigational Sites, Bogen
  - Teva Investigational Sites, Bonn
  - Teva Investigational Sites, Butzbach
  - Teva Investigational Sites, Buxtehude
  - Teva Investigational Sites, Chemnitz
  - Teva Investigational Sites, Cloppenburg
  - Teva Investigational Sites, Cologne
  - Teva Investigational Sites, Cottbus
  - Teva Investigational Sites, Dessau
  - Teva Investigational Sites, Dillingen
  - Teva Investigational Sites, Düsseldorf
  - Teva Investigational Sites, Eisleben Lutherstadt
  - Teva Investigational Sites, Erbach im Odenwald
  - Teva Investigational Sites, Erfurt
  - Teva Investigational Sites, Essen
  - Teva Investigational Sites, Flensburg
  - Teva Investigational Sites, Frankfurt
  - Teva Investigational Sites, Fürth
  - Teva Investigational Sites, Gadebusch
  - Teva Investigational Sites, Gelsenkirchen
  - Teva Investigational Sites, Gera
  - Teva Investigational Sites, Gladenbach
  - Teva Investigational Sites, Göppingen
  - Teva Investigational Sites, Göttingen
  - Teva Investigational Sites, Greifswald
  - Teva Investigational Sites, Großbeeren
  - Teva Investigational Sites, Grünstadt
  - Teva Investigational Sites, Hagen
  - Teva Investigational Sites, Halsbrücke
  - Teva Investigational Sites, Hamburg
  - Teva Investigational Sites, Hanover
  - Teva Investigational Sites, Heidenheim
  - Teva Investigational Sites, Herne
  - Teva Investigational Sites, Hettstedt
  - Teva Investigational Sites, Hildesheim
  - Teva Investigational Sites, Hoppegarten
  - Teva Investigational Sites, Ilmenau
  - Teva Investigational Sites, Immenstadt im Allgäu
  - Teva Investigational Sites, Iserlohn
  - Teva Investigational Sites, Itzehoe
  - Teva Investigational Sites, Jülich
  - Teva Investigational Sites, Kaiserslautern
  - Teva Investigational Sites, Karlstadt am Main
  - Teva Investigational Sites, Kastellaun
  - Teva Investigational Sites, Katzenelnbogen
  - Teva Investigational Sites, Kaufbeuren
  - Teva Investigational Sites, Kempten
  - Teva Investigational Sites, Kiel
  - Teva Investigational Sites, Kleve
  - Teva Investigational Sites, Königsbrück
  - Teva Investigational Sites, Krefeld
  - Teva Investigational Sites, Ladenburg
  - Teva Investigational Sites, Landshut
  - Teva Investigational Sites, Lappersdorg
  - Teva Investigational Sites, Lauf
  - Teva Investigational Sites, Leer
  - Teva Investigational Sites, Leipzig
  - Teva Investigational Sites, Leverkusen
  - Teva Investigational Sites, Limburg
  - Teva Investigational Sites, Lingen
  - Teva Investigational Sites, Lohr
  - Teva Investigational Sites, Ludwigshafen
  - Teva Investigational Sites, Magdeburg
  - Teva Investigational Sites, Mainz
  - Teva Investigational Sites, Mannheim
  - Teva Investigational Sites, Markkleeberg
  - Teva Investigational Sites, Menden
  - Teva Investigational Sites, Mittweida
  - Teva Investigational Sites, Mönchengladbach
  - Teva Investigational Sites, Mühlhausen
  - Teva Investigational Sites, München
  - Teva Investigational Sites, Naumburg
  - Teva Investigational Sites, Neu-Ulm
  - Teva Investigational Sites, Neuburg am Inn
  - Teva Investigational Sites, Neunkirchen
  - Teva Investigational Sites, Neupotz
  - Teva Investigational Sites, Neusäß
  - Teva Investigational Sites, Nuremberg
  - Teva Investigational Sites, Oberhausen
  - Teva Investigational Sites, Oldenburg
  - Teva Investigational Sites, Osnabrück
  - Teva Investigational Sites, Ostfildern
  - Teva Investigational Sites, Pulheim
  - Teva Investigational Sites, Ravensburg
  - Teva Investigational Sites, Regensburg
  - Teva Investigational Sites, Ribnitz-Damgarten
  - Teva Investigational Sites, Rostock
  - Teva Investigational Sites, Rotenburg (Wümme)
  - Teva Investigational Sites, Saalouis
  - Teva Investigational Sites, Sande
  - Teva Investigational Sites, Schirgiswalkde-Kirschau
  - Teva Investigational Sites, Schleiden
  - Teva Investigational Sites, Schongau
  - Teva Investigational Sites, Schwarzenbruck
  - Teva Investigational Sites, Schweich
  - Teva Investigational Sites, Schweinfurt
  - Teva Investigational Sites, Schwerin
  - Teva Investigational Sites, Schwetzingen
  - Teva Investigational Sites, Seelow
  - Teva Investigational Sites, Siegen
  - Teva Investigational Sites, Sinsheim
  - Teva Investigational Sites, Solingen
  - Teva Investigational Sites, Sondershausen
  - Teva Investigational Sites, Sprockhövel
  - Teva Investigational Sites, Stade
  - Teva Investigational Sites, Stralsund
  - Teva Investigational Sites, Stuttgart
  - Teva Investigational Sites, Treuenbrietzen
  - Teva Investigational Sites, Troisdorg-Sieglar
  - Teva Investigational Sites, Tübingen
  - Teva Investigational Sites, Ulm
  - Teva Investigational Sites, Varel
  - Teva Investigational Sites, Vellmar
  - Teva Investigational Sites, Weißenfels
  - Teva Investigational Sites, Wismar
  - Teva Investigational Sites, Wolfach
  - Teva Investigational Sites, Wolfratshausen
  - Teva Investigational Sites, Wuppertal
  - Teva Investigational Sites, Zossen
  - Teva Investigational Sites, Zwickau